CLINICAL TRIAL: NCT00078910
Title: A Prospective Phase II Study of Preoperative, Controlled Exisulind Therapy Initiated Prior to Radical Prostatectomy: Effect on Apoptosis
Brief Title: Neoadjuvant Exisulind in Treating Patients Who Are Undergoing Radical Prostatectomy for Stage II or Stage III Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Purpose: Treatment
Other Study IDs: CDR0000353196; MAYO-229701
Record Dates: First submitted 2004-03-08; First posted 2004-03-09 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2006-09

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — sulindac sulfone; Neoadjuvant Therapy

INTERVENTIONS:
Drug: exisulind
Procedure: conventional surgery
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as exisulind, work in different ways to stop tumor cells from dividing so they stop growing or die. Giving a chemotherapy drug before surgery may shrink the tumor so that it can be removed.

PURPOSE: This phase II trial is studying how well neoadjuvant exisulind works in treating patients who are undergoing radical prostatectomy for stage II or stage III prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the effect of neoadjuvant exisulind vs no neoadjuvant treatment on apoptosis in patients with stage II or III prostate cancer undergoing radical prostatectomy.

Secondary

* Determine the effect of this drug (preoperatively) on surrogate endpoint biomarkers (i.e., prostate-specific antigen, high-grade prostatic intraepithelial neoplasia, MIB-1, and DNA ploidy) in these patients.

OUTLINE: This is a nonrandomized, controlled study. Patients are assigned to 1 of 2 groups based on the treating physician.

* Control group: Patients undergo radical prostatectomy only.
* Treatment group: Patients receive oral exisulind once daily for 4 weeks. Patients then undergo radical prostatectomy.

Patients are followed at 1 month.

PROJECTED ACCRUAL: A total of 130 patients (65 per group) will be accrued for this study within approximately 10-12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * Clinical stage T1c-3b, N0-X, M0
  * Gleason score ≥ 6
* Planning to undergo pelvic lymphadenectomy and radical prostatectomy at Mayo Clinic Rochester

  * Interval from biopsy to prostatectomy is at least 4, but no more than 14, weeks
  * Selected patients of Dr. R. P. Myers who are undergoing prostatectomy during the enrollment period will be assigned to the control group* NOTE: *Additional historical controls may be selected from Dr. Myers' patients who underwent prostatectomy within the past 4 years

PATIENT CHARACTERISTICS:

Age

* 40 and over

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* ALT normal (10-45 U/L)
* AST normal (12-31 U/L)
* Alkaline phosphatase normal (119-309 U/L)
* Bilirubin normal (0.1-1.0 mg/dL)
* No history of hepatitis, cirrhosis, or other hepatic dysfunction

Renal

* Creatinine < 1.5 mg/dL

Other

* Fertile patients must use effective contraception
* No hypersensitivity to sulindac (treatment group)

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent immunotherapy

Chemotherapy

* No other concurrent chemotherapy

Endocrine therapy

* No prior ablation (treatment group)
* No prior hormone replacement or antiandrogen therapy (e.g., testosterone, diethylstilbestrol, leuprolide, goserelin, flutamide, bicalutamide, finasteride, nilutamide, or megestrol)
* No concurrent antiandrogen therapy, luteinizing hormone-releasing hormone agonists, finasteride, or diethylstilbestrol

Radiotherapy

* No prior pelvic radiotherapy
* No concurrent radiotherapy

Surgery

* See Disease Characteristics

Other

* No prior treatment for prostate cancer before prostatectomy (control group)
* No concurrent cyclooxygenase-2 inhibitors
* No concurrent sulindac
* No concurrent nonsteroidal anti-inflammatory drugs except low-dose (no more than 325 mg/day) aspirin for cardiovascular prophylaxis

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2003-08; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Apoptosis 4 weeks after completion of study as assessed by marker analysis (bcl-2, Bax, Par-4, M30, TUNEL assay, PTEN)

SECONDARY OUTCOMES:
Modulation of other surrogate endpoint biomarkers (prostate-specific antigen high-grade prostatic intraepithelial neoplasia, MIB-1, and DNA ploidy)

CONTACTS AND LOCATIONS:
Overall Officials: Bradley C. Leibovich, MD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Mayo Clinic Cancer Center, Rochester, Minnesota